CLINICAL TRIAL: NCT06733961
Title: Investigation of the Relationship of SCUBE-1 and VAP-1 Levels on Diagnosis, Prognosis and Clinical Results in Patients with Pulmonary Thromboembolism Diagnosis in Emergency Department
Brief Title: SCUBE-1 and VAP-1 Levels on Diagnosis Pulmonary Embolism
Status: Completed | Type: Observational
Sponsor: Giresun University (Other)
Responsible Party: Principal Investigator, İskender Aksoy, Assistant Professor, Giresun University
Other Study IDs: OMÜ KAEK 2019/26
Record Dates: First submitted 2024-12-01; First posted 2024-12-13 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-11

CONDITIONS: Pulmonary Embolism Acute
Keywords: SCUBE-1; VAP-1; Pulmonary Embolism
MeSH Terms: conditions — Pulmonary Embolism

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples Without DNA — To study SCUBE-1 and VAP-1, 5 cc of blood was taken from each patient and healthy volunteer.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patient group: It consists of patients diagnosed with Pulmonary Thromboembolism who meet the inclusion and exclusion criteria.
  Interventions: Diagnostic Test: SCUBE-1 and VAP-1
- Control group: It was composed of healthy volunteers of similar age and gender who did not have any acute complaints.
  Interventions: Diagnostic Test: SCUBE-1 and VAP-1

INTERVENTIONS:
Diagnostic Test: SCUBE-1 and VAP-1 — There is no other study comparing these biomarkers with healthy volunteers in the diagnosis of pulmonary embolism.

SUMMARY:
Acute pulmonary thromboembolism is a life-threatening disease. Clinical suspicion is essential for diagnosis because of lack of a specific finding for diagnosis of PTE. The aim of this study is to investigate the relationship between the diagnosis and prognosis of alternative biomarkers such as SCUBE-1 and VAP-1 in the diagnosis of clinically suspected acute PTE.

Patients who were admitted to the Emergency Department and diagnosed as acute PTE were included in the study. Patients with acute ischemic disease, liver failure, renal failure, pregnancy, active malignancy and/or history of known PTE were excluded from the study. A control group was formed from healthy volunteers at similar age and sex. SCUBE-1 and VAP-1 levels were studied from serum samples taken from the patient and control groups. Data were analyzed using by IBM SPSS V23.

DETAILED DESCRIPTION:
The definitive diagnosis of APT is made by ventilation/perfusion (V/Q) scintigraphy and thorax computed tomography angiography (CTA). There is no specific examination as a laboratory parameter. A definitive diagnosis cannot be made with d-Dimer, which is the most frequently used laboratory test today; it is used to exclude the diagnosis of APT.

The non-specificity of the clinical picture, the fact that the diagnosis depends on the experience of the physician and the necessity of exposure to radiation and contrast material for the definitive diagnosis has revealed the necessity of searching for alternative ways for the diagnosis of APT. "Signal peptide CUB-EGF domain-containing protein-1" (SCUBE-1) is a biomarker released during platelet aggregation, and "Vascular adhesion protein-1" (VAP-1) is a biomarker released from endothelium, and these biomarkers show promise for the diagnosis of APT.

Determination of serum SCUBE-1 and serum VAP-1 levels 5 mL blood taken from the peripheral veins of the patients was placed in a biochemistry tube and centrifuged at 3000 g. After centrifugation, the serum part of the blood was separated and taken into an eppendorf tube and stored in an ultra-deep freezer at minus 80°C until the study day. Before starting the study, the ELISA kits kept at 2-8°C and the samples kept in an ultra-deep freezer at minus 80°C were brought to room temperature.

ELIGIBILITY:
Inclusion Criteria:

* being older than 18 years of age
* presenting to the emergency department,
* diagnosed with acute PTE by contrast-enhanced computed tomography angiography

Exclusion Criteria:

* having acute ischemic disease, liver, kidney or advanced heart failure, liver disease, pregnancy, active malignancy or hematological disease, and a known history of PTE.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who applied to the emergency department of Samsun Ondokuz Mayis Universtiy between 01.01.2019 and 30.06.2019 and were diagnosed with acute pulmonary thromboembolism (APT) by contrast-enhanced thorax computed tomography were included in the study. A group of healthy volunteers with similar gender, age and exclusion criteria was formed with the patients with APT included in the study. Demographic data, clinical probability scores (Wells' criteria, revised Geneva score), simplified Pulmonary Embolism Severity Index (sPESI) and early mortality risk score (in 30 days) of the patients were recorded.
Sampling Method: Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Diagnostic ability of SCUBE-1 and VAP-1 in pulmonary embolism | 6 month
  Serum SCUBE-1 and serum VAP-1 levels of the Patient and Control groups will be measured in serum mg/dL with 5 mL of blood taken from the peripheral veins.

SECONDARY OUTCOMES:
Difference between clinical probability scores and serum SCUBE-1 and VAP-1 levels. | 6 month
  The clinical probability scores of the patient group will be grouped as 'low, medium, high' and 'APT likely, APT unlikely'. Serum SCUBE-1 and serum VAP-1 levels measured in the patient group will be measured in the subgroups of clinical probability scores.
difference between early mortality risk and serum SCUBE-1 and VAP-1 levels. | 28 days
  For the patient group, 'low, medium-low, medium-high, high' risk groups will be determined for the 28-day early mortality risk. Serum SCUBE-1 and serum VAP-1 levels will be measured for these subgroups.

CONTACTS AND LOCATIONS:
Overall Officials: Hizir U. Akdemir, Prof., Study Chair — Ondokuz Mayıs University
Locations (1):
- Ondokuz Mayis University, Samsun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dirican N, Duman A, Saglam G, Arslan A, Ozturk O, Atalay S, Bircan A, Akkaya A, Cakir M. The diagnostic significance of signal peptide-complement C1r/C1s, Uegf, and Bmp1-epidermal growth factor domain-containing protein-1 levels in pulmonary embolism. Ann Thorac Med. 2016 Oct-Dec;11(4):277-282. doi: 10.4103/1817-1737.191876. PMID 27803754
- [Background] Turkmen S, Sahin A, Gunaydin M, Sahin S, Mentese A, Turedi S, Karahan SC, Ozsu S, Gunduz A. The value of signal peptide-CUB-EGF domain-containing protein-1 (SCUBE1) in the diagnosis of pulmonary embolism: a preliminary study. Acad Emerg Med. 2015 Aug;22(8):922-6. doi: 10.1111/acem.12721. Epub 2015 Jul 22. PMID 26202675